CLINICAL TRIAL: NCT06489093
Title: Evaluation of the Effect of Green Synthesized Nano-silver Fluoride and Silver Diamine Fluoride on Carious Lesions in Children
Brief Title: Remineralizing Effect of Different Silver-containing Agents on Initial Caries Lesions in Primary Teeth in Children
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-841/08.04.2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: White Spot Lesion of Tooth
Keywords: sdf; nano silver fluoride; white spot lesions
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NSF (Gr-N) (Experimental): The Gr-N will receive treatment with green synthesized Nano silver fluoride which is laboratory conducted
  Interventions: Drug: NSF
- SDF+KI group (Gr-S) (Active Comparator): The Gr-S will receive treatment with SDF + KI (Riva Star 38% , SDI) according to the manufacturer's instructions.
  Interventions: Drug: SDF+KI
- Control group (Gr-C) (Placebo Comparator): The control group (Gr-C) receive no intervention except brushing twice daily with aminofluoride toothpaste and toothbrush provided by researcher.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: NSF — Prior to treatment the working field is isolated with cotton rolls. Gingival barrier is used for soft tissue protection. Application of NSF using a microapplicator on the carious lesion for 1 minute. Excess material and gingival barrier are removed. Participants receive oral hygiene instructions.
  Other Names: green synthesized Nano silver fluoride
  Arms: NSF (Gr-N)
Drug: SDF+KI — Prior to treatment the working field is isolated with cotton rolls. Gingival barrier is used for soft tissue protection. Application of 38% silver diamine fluoride (Riva star 38%, SDI) using a microapplicator on the carious lesion. Immediately afterwards, potassium iodide is applied as a reducing agent. Excess material and gingival barrier are removed. Participants receive oral hygiene instructions.
  Other Names: Riva star 38%, SDI
  Arms: SDF+KI group (Gr-S)
Other: Control group — Subjects will receive oral hygiene instructioins to apply fluoridated toothpaste to a toothbrush and brush teeth thoroughly for at least 2 minutes, then expectorate and rinse.
  Arms: Control group (Gr-C)

SUMMARY:
The aim of the present work is to study the effect of the application of Silver diamine fluoride (SDF) and a novel green synthesized Nano-silver fluoride (NSF) on early enamel lesions in primary teeth. Proving their positive effect would be the basis for the development of innovative dental materials and hygienic agents to combat the carious process, which is a critical prerequisite for improving the quality of dental services and reducing dental anxiety and fear.

DETAILED DESCRIPTION:
Dental caries is a major public health concern, especially in very young children. Early detection of the disease enhances and simplifies treatment effectiveness. Non-operative treatments are particularly advantageous as they are minimally invasive, reduce future operative treatment needs and are more comfortable, thereby improving overall compliance and dental experience.

The aim of the study is to compare the clinical efficacy of Silver diamine fluoride (SDF) and laboratory prepared green synthesized Nano-silver fluoride on early enamel lesions in primary teeth.

The proposed study is a randomized controlled clinical trial. Included patients are healthy positive children aged from 3 to 8 years, requiring non-operative treatment of incipient caries lesions on smooth surfaces of primary teeth. Lesions will be assessed visually using ICDAS II, Nyvad criteria and laser fluorescence (LF pen).

Patients are randomly assigned to one of three study groups:

Group N: Green synthesized Nano silver fluoride (prepared in laboratory) Group S: SDF + KI (38% Riva Star, SDI) Group C: Control group

Prior to treatment parents are informed about the nature of the study and sign an informed consent. Children are introduced to the method of conducting treatment in a style appropriate for the child's age. Lesions are assesed using the ICDAS II system, Nyvad criteria and laser fluorescence. All patients receive professional oral hygiene with a fluoride-free brush and polishing paste. Treatment of each patient's respective teeth is performed following the treatment protocol of the respective agents. Follow-ups are performed at 1st, 3rd, 6th and 12th month.

ELIGIBILITY:
Inclusion Criteria:

* Age: 3 - 8 years
* Signed informed consent from parents to participate in the study. Verbal consent from the child for the upcoming manipulations.
* Enrolled patients do not have any common diseases or conditions associated with decreased salivation and are not taking medications that suppress salivary flow. Study participants have no cognitive or behavioral impairment. The absence of disease will be confirmed by a history-taking interview with the parent.
* Presence of incipient carious lesions (white spots) reaching the enamel interior, assessed with ICDAS system values 01 (first visible enamel change) and 02 (localized visible enamel change) and laser fluorescence values up to 20. The diagnostic threshold of the included lesions is defined as D1 A (active enamel lesion visible after drying) or D2 A (active enamel lesion visible without drying). Criteria for active lesions: under plaque, loss of gloss, loss of smoothness, diffuse borders of the lesion, opaque appearance, white colour, at pre-selection sites (in the cervical third of the enamel). The lesions are located on tooth surfaces with no preceding obturations.
* Study participants had not performed remineralization or topical fluoride therapy on the included lesions within six months prior to study inclusion.
* Children with no history of allergy to the medications administered.

Exclusion Criteria:

* Children who are considered medically compromised or medically complex patients. The presence of a medical condition is confirmed by a history interview with the child's parent or guardian and involves common diseases or conditions associated with decreased salivation and intake of medications that suppress salivary flow, cognitive and behavioral disorders.
* Patients who underwent remineralizing or topical fluoride therapy to the included lesions in the last six months prior to study inclusion.
* Patients with a history of allergy to the administered medication.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-07-29 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Visual assessment using ICDAS II coding system | 12 months (Baseline, 1 month, 3 months, 6 months and 12 months)
  Code 0: Sound tooth surface Code 1: First visual change in enamel. Code 2: Distinct visual change in enamel visible when wet, lesion must be visible when dry.
  Code 3: Localized enamel breakdown because of caries with no visible dentin or underlying shadow.
  Code 4: Underlying dark shadow from dentin with or without localized enamel breakdown.
  Code 5: Distinct cavity with visible dentin. Code 6: Extensive distinct cavity with visible dentin.
  After treatment, the evaluation will be performed as follows: Increase to ICDAS 3 or more indicates caries progression; decrease to 0-1 this indicates caries regression. If score remains the same this indicates no change in lesion.
  No. of lesions with scores 0,1,2,3 or more will be assessed and analyzed.
Activity of a carious lesion using Nyvad Caries Diagnostic Criteria | 12 months (Baseline, 1 month, 3 months, 6 months and 12 months)
  Code 0: Sound (normal) enamel Code 1: Active caries (intact surface) - Surface of enamel is whitish/yellowish opaque Code 2: Active caries (surface discontinuity) Code 3: Active caries (cavity) - Enamel/dentin cavity easily visible with the naked eye.
  Code 4: Inactive caries (intact surface) - Surface of enamel is whitish, brownish or black.
  Code 5: Inactive caries (surface discontinuity) - Same criteria as score 4. Localized surface defect (microcavity) in enamel only Code 6: Inactive caries (cavity) - Enamel/dentin cavity easily visible with the naked eye; surface of cavity may be shiny and feels hard on probing with gentle pressure.
  Code 7: Filling (sound surface) Code 8: Filling + active caries - Caries lesion may be cavitated or noncavitated.
  Code 9: Filling + inactive caries - Caries lesion may be cavitated or noncavitated.
Change in lesion fluorescence evaluated using diode laser fluorescence device | 12 months (Baseline, 1 month, 3 months, 6 months and 12 months)
  Laser fluorescence values are categorized using the following scale:
  0-5 - no change 5-10 - enamel caries located in the outer enamel surface 10-15 - enamel caries located to the middle of the enamel 15-20 - enamel caries reaching the dentine enamel junction >20 - caries in the dentine

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Palankalieva, DMD, Principal Investigator — Department Of Pediatric Dentistry, Faculty Of Dental Medicine, Medical University Of Plovdiv, Bulgaria
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dental Medicine, Medical University-Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No